CLINICAL TRIAL: NCT03657095
Title: An Open-label Extension of BPS-314d-MR-PAH-302 in Pulmonary Arterial Hypertension Patients
Brief Title: A Study With BPS-314d-MR-PAH-303 in Participants With Pulmonary Arterial Hypertension
Acronym: BEAT OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The pivotal study, BPS-314d-MR-PAH-302 (NCT01908699), failed to demonstrate efficacy.
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPS-314d-MR-PAH-303
Record Dates: First submitted 2018-05-18; First posted 2018-09-04 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Hypertension; Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Lung Diseases; Vascular Diseases; Cardiovascular Diseases; Respiratory Tract Diseases; Prostacyclin; Beraprost; Epoprostenol; Platelet Aggregation Inhibitors; Vasodilator Agents; Antihypertensive Agents
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension; Familial Primary Pulmonary Hypertension; Hypertension, Pulmonary; Lung Diseases; Vascular Diseases; Cardiovascular Diseases; Respiratory Tract Diseases | interventions — beraprost

STUDY DESIGN:
Masking Description: Treatment during the first 4 weeks of this study will be double-blind. The Investigator and study staff, the participants, the monitors, and the Sponsor will remain blinded to the treatment group allocation from BPS-314d-MR-PAH-302 double-blind study (NCT01908699) and to study drug during the first 4 weeks of the OLE study while the participants transition to the OLE treatment. After the 4 weeks, the study will continue as unblinded and open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Esuberaprost (Experimental): Participants who received esuberaprost during the BPS-314d-MR-PAH-302 double-blind study will receive 2 tablets of 15 μg esuberaprost sodium tablets for oral administration QID for up to 7 months (which will include the 4 weeks of blinded transition).
  Interventions: Drug: Esuberaprost
- Placebo/Esuberaprost (Placebo Comparator): Participants who received placebo during the BPS-314d-MR-PAH-302 double-blind study will receive 1 esuberaprost tablet and 1 placebo tablet QID during the first 2 weeks of the blinded transition and then receive 2 esuberaprost tablets QID for the rest of the study, for up to 7 months (which will include the other 2 weeks of the total 4-week blinded transition).
  Interventions: Drug: Esuberaprost; Drug: Placebo

INTERVENTIONS:
Drug: Esuberaprost — Sodium tablets
  Other Names: Beraprost Sodium 314d Modified Release tablets
Drug: Placebo — Placebo tablets, which are identical in size and appearance to those containing Esuberaprost.
  Arms: Placebo/Esuberaprost

SUMMARY:
This is a multi-center, open-label study for eligible participants who were actively participating in the BPS-314d-MR-PAH-302 double-blind study (NCT01908699) at the time the study was concluded. This open-label extension (OLE) study will evaluate the safety, tolerability, and efficacy of long-term treatment with esuberaprost sodium tablets (Beraprost Sodium 314d Modified Release tablets).

DETAILED DESCRIPTION:
Participants will sign an informed consent to continue treatment for pulmonary arterial hypertension (PAH) with esuberaprost sodium tablets in this OLE study. At the Enrollment Visit for this OLE study, participants will begin a blinded transition from the BPS-314d-MR-PAH-302 double-blind study to this study over 4 weeks. The first dose for all participants in this OLE study will be 2 tablets. During this blinded transition, those participants on active study drug in the BPS-314d-MR-PAH-302 study will continue with blinded active study drug 4-times daily (QID); those participants who were on placebo study drug will receive 1 active tablet and 1 placebo tablet QID (blinded) during the first 2 weeks and increase to 2 active tablets QID (blinded) thereafter. After the first dose, the Investigator may adjust the dose as medically warranted. The maximum dose for this study is 30 microgram (μg) QID with a minimum accepted dose as 15 μg QID. For the first 4 weeks, contact with the participant should occur weekly to ensure up-titration to the fixed dose is tolerated and assess adverse events (AEs).

Participants will return to the clinic at Week 4 to be supplied open-label esuberaprost sodium tablets and complete protocol specified procedures. At the Week 4 Visit, participants will be dosed with two 15 μg tablets (30 μg total), administered orally QID (provided the target dose is tolerated), or follow the Investigator's (or designee's) directions if adjustment is needed. Following the Week 4 Visit, each participant will return to the clinic at Months 3, 6, 9, and 12, and quarterly thereafter for assessments.

This study is expected to continue until the first of any of the following are reached: the study drug is commercially available, the Sponsor discontinues the study, or the Sponsor offers enrollment in another study (estimated to be up to 2 years). At the conclusion of the study or if a participant discontinues the study prematurely, participants will return to the clinic for an End-of-Study (EOS) Visit. Participants will be provided instructions about down titration off esuberaprost sodium tablets by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have been actively participating in the double-blind study, BPS-314d-MR-PAH-302 (NCT01908699), when the Sponsor concluded that study.
2. In the Investigator's opinion, participant must be competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved informed consent form (ICF) and must sign the form prior to the initiation of any study procedures.
3. Women of child-bearing potential (defined as less than 1 year post-menopausal and not surgically sterile) must be practicing abstinence or using 2 highly-effective methods of contraception (defined as a method of birth control that results in a low failure rate [that is, less than 1% per year, such as approved hormonal contraceptives, barrier methods (such as a condom or diaphragm) used with a spermicide or an intrauterine device]). Participant must have a negative pregnancy test at the BPS-314d-MR-PAH-302 EOS Visit / BPS-314d-MR-PAH-303 Enrollment Visit.
4. Participant must be willing and able to comply with study requirements and restrictions.

Exclusion Criteria:

1. Participant is pregnant or lactating.
2. Participant is scheduled to receive another investigational drug, device, or therapy during the course of the study.
3. Participant is taking or intends to take any prostacyclin / prostacyclin (IP) analog or IP receptor agonist (except for treprostinil, inhaled [Tyvaso®]).
4. Participant has any other clinically significant illness or other reason that, in the opinion of the Investigator, might put the participant at risk of harm during the study or might adversely affect the interpretation of the study data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (43):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - University of California San Diego Medical Center, La Jolla, California
  - University of California Los Angeles UCLA, Los Angeles, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - Santa Barbara Pulmonary Associates, Santa Barbara, California
  - Stanford Hospital and Clinics, Stanford, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Allianz Research Institute, Westminster, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Bay Area Cardiology Research, Brandon, Florida
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - South Miami Heart Specialists, South Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Georgia Clinical Research, Austell, Georgia
  - Indiana University Health North Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beaumont Health, Troy, Michigan
  - Albany Medical Center, Albany, New York
  - The Mount Sinai Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The University of Toledo, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Anderson Pharmaceutical Research, LLC, Anderson, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the Enrollment Visit for this open-label extension (OLE) study, participants began a blinded transition from the pivotal BPS-314d-MR-PAH-302 double-blind study (NCT01908699) to this study over 4 weeks.
Groups:
- Esuberaprost: Participants who received esuberaprost during the BPS-314d-MR-PAH-302 double-blind study received 2 tablets of 15 microgram (μg) esuberaprost sodium tablets for oral administration 4 times daily (QID) for up to 7 months (which included the 4 weeks of blinded transition).
- Placebo/Esuberaprost: Participants who received placebo during the BPS-314d-MR-PAH-302 double-blind study received 1 esuberaprost tablet and 1 placebo tablet QID for the first 2 weeks of the blinded transition and then received 2 esuberaprost tablets QID for the rest of the study, for up to 7 months (which included the other 2 weeks of the total 4-week blinded transition).
Period: Overall Study
Arm/Group | Esuberaprost | Placebo/Esuberaprost
Started | 59 | 53
Received at Least 1 Dose of Study Drug | 59 | 53
Completed | 0 | 0
Not Completed | 59 | 53
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Study Terminated by Sponsor | 58 | 49

BASELINE CHARACTERISTICS:
Population: All participants who receive at least 1 dose of study drug.
Groups:
- Esuberaprost: Participants who received esuberaprost during the BPS-314d-MR-PAH-302 double-blind study received 2 tablets of 15 μg esuberaprost sodium tablets for oral administration QID for up to 7 months (which included the 4 weeks of blinded transition).
- Total: Total of all reporting groups
Arm/Group | Esuberaprost | Placebo/Esuberaprost | Total
Number analyzed (Participants) | 59 | 53 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.02) | 62.5 (9.75) | 60.6 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 53 | 49 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 9 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 49 | 44 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is any untoward medical occurrence or undesirable event(s) experienced in a participant that begins or worsens following administration of study drug, whether or not considered related to study drug by Investigator. A serious adverse event (SAE) is an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason, death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), or persistent or significant disability/incapacity. AEs included both SAEs and non-serious AEs. AEs were coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Month 7
Population: All participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Esuberaprost | Placebo/Esuberaprost
Number analyzed (Participants) | 59 | 53
Participants
  TEAEs | 56 | 52
  Treatment-Emergent SAEs | 9 | 8

2. Secondary Outcome: Area Walked for the 6 Minute Walk Distance (6MWD) Test
Description: Area used for the Six Minute Walk Test (6MWT) were to be pre-measured at 30 meters in length. Rest periods were to be allowed if participant could no longer continue. If participant needed to rest, he/she could have stood or sit and then begin again when rested but the clock would continue to run. At the end of 6 minutes, the tester was to call "stop" while stopping the watch and then measure the distance walked. Distance <500 meters would have suggested considerable exercise limitation; distance 500-800 meters would have suggested moderate limitation; and distance >800 meters (with no rests) would have suggested mild or no limitation. This extension study was terminated early due to the pivotal double-blind study failed to demonstrate efficacy. Therefore, efficacy data was not collected or analyzed.
Time Frame: Week 4 and then every 3 months until study termination (Month 7)
Population: All participants who receive at least 1 dose of study drug. Efficacy data was not collected or analyzed for this extension study.
Arm/Group | Esuberaprost | Placebo/Esuberaprost
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Borg Dyspnea Score
Description: The modified 0-10 category-ratio Borg scale is one in which the participants were to rate the maximum level of dyspnea they experienced during the 6MWT. Scores would have ranged from 0 (for the best condition) and 10 (for the worst condition). This extension study was terminated early due to the pivotal double-blind study failed to demonstrate efficacy. Therefore, efficacy data was not collected or analyzed. Note, a summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Week 4 and then every 3 months until study termination (Month 7)
Population: as for outcome 2
Arm/Group | Esuberaprost | Placebo/Esuberaprost
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants in Each Category of the World Health Organization (WHO) Functional Class (FC)
Description: The WHO Functional Class of pulmonary hypertension is a physical activity rating scale as follows: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms. This extension study was terminated early due to the pivotal double-blind study failed to demonstrate efficacy. Therefore, efficacy data was not collected or analyzed.
Time Frame: Week 4 and then every 3 months until study termination (Month 7)
Population: as for outcome 2
Arm/Group | Esuberaprost | Placebo/Esuberaprost
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With a TEAE of N-terminal Pro-brain Natriuretic Peptide (NT-pro-BNP) Increased
Description: A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Month 7
Population: All participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Esuberaprost | Placebo/Esuberaprost
Number analyzed (Participants) | 59 | 53
Participants | 5 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Month 7
Description: Adverse events were collected from all participants who receive at least 1 dose of study drug.
Arm/Group | Esuberaprost | Placebo/Esuberaprost
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/53
Serious Adverse Events (participants affected / at risk) | 12/59 | 8/53
Other Adverse Events (participants affected / at risk) | 56/59 | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esuberaprost (N=59) | Placebo/Esuberaprost (N=53)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1
Coronary artery compression (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Esuberaprost (N=59) | Placebo/Esuberaprost (N=53)
Diarrhoea (Gastrointestinal disorders) | 9 | 12
Nausea (Gastrointestinal disorders) | 7 | 8
Constipation (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Glossitis (Gastrointestinal disorders) | 2 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Mucous stools (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 21 | 17
Dizziness (Nervous system disorders) | 9 | 9
Disturbance in attention (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Amputation stump pain (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Sclerodactylia (Musculoskeletal and connective tissue disorders) | 1 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 9 | 9
Oedema peripheral (General disorders) | 7 | 6
Chest discomfort (General disorders) | 4 | 3
Pain (General disorders) | 1 | 4
Peripheral swelling (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 1
Oedema (General disorders) | 2 | 0
Calcinosis (General disorders) | 1 | 0
Crepitations (General disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 0 | 1
Feeling cold (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 4 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3
Pneumonia (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 2 | 0
Herpes virus infection (Infections and infestations) | 2 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Helminthic infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Nasal vestibulitis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 5 | 2
Weight increased (Investigations) | 4 | 2
Blood creatinine increased (Investigations) | 2 | 2
Blood urea increased (Investigations) | 3 | 1
Blood uric acid increased (Investigations) | 3 | 1
Haemoglobin decreased (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Electrocardiogram T wave inversion (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Haematocrit increased (Investigations) | 1 | 1
Haemoglobin increased (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Antinuclear antibody positive (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood HIV RNA increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood iron decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0
Carbon dioxide decreased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Heart sounds abnormal (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Protein urine (Investigations) | 1 | 0
Prothrombin time abnormal (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
QRS axis abnormal (Investigations) | 1 | 0
Serum ferritin decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Flushing (Vascular disorders) | 9 | 3
Hot flush (Vascular disorders) | 2 | 4
Hypertension (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1
Palpitations (Cardiac disorders) | 6 | 3
Bradycardia (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery compression (Cardiac disorders) | 1 | 0
Coronary ostial stenosis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 3 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Polycythaemia (Blood and lymphatic system disorders) | 2 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Dry eye (Eye disorders) | 1 | 1
Eye irritation (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seasonal allergy (Immune system disorders) | 3 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hypercalciuria (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Hypocitraturia (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/16 | 1/14 — This is a sex-specific adverse event that only affects male participants.
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0/43 | 1/39 — This is a sex-specific adverse event that only affects female participants.
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1/43 | 0/39 — This is a sex-specific adverse event that only affects female participants.
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Tornwaldt cyst (Congenital, familial and genetic disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to the pivotal study, BPS-314d-MR-PAH-302 (NCT01908699), failed to demonstrate efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT03657095/Prot_SAP_001.pdf